CLINICAL TRIAL: NCT00157924
Title: A Multicenter, Randomized, Open-label Study to Evaluate the Lipid-Altering Efficacy and Safety of Ezetimibe (+) Simvastatin Versus Atorvastatin in Hypercholesterolemic Patients With Diabetes Mellitus or Metabolic Syndrome
Brief Title: Ezetimibe (+) Simvastatin vs. Atorvastatin Comparative Study in DM or Metabolic Syndrome Patients (0653A-093)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-093; MK0653A-093; 2005_064
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

ARMS (2):
- 1 (Experimental): 1. simvastatin/ezetimibe 10/20mg
  Interventions: Drug: simvastatin (+) ezetimibe
- 2 (Active Comparator): 2. atorvastatin 10mg
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: simvastatin (+) ezetimibe — simvastatin (+) ezetimibe 10/20mg.
  Other Names: MK0653A; Vytorin®
  Arms: 1
Drug: atorvastatin — atorvastatin 10mg
  Other Names: Lipitor®
  Arms: 2

SUMMARY:
An efficacy and safety study of ezetimibe (+) simvastatin compared to atorvastatin at week 6 in diabetics or metabolic syndrome patients in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypercholesterolemia
* Drug naive or statin treated but inadequately controlled patients against NCEP ATP III guideline goal

Exclusion Criteria:

* Hypersensitivity to HMG-CoA inhibitor or Ezetimibe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
LDL-C lowering efficacy | 6 weeks

SECONDARY OUTCOMES:
Safety | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html